CLINICAL TRIAL: NCT05878340
Title: "Miffy Eats the Rainbow!" Efficiency of Stimulating Colour Consumption as Strategy to Increase Fruit and Vegetable Intake in Children
Brief Title: Miffy Eats the Rainbow
Acronym: Miffy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wageningen University (Other)
Responsible Party: Principal Investigator, Guido Camps, Principal investigator, Wageningen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: Miffy Study
Record Dates: First submitted 2023-04-25; First posted 2023-05-26 (Actual); Last update posted 2023-05-26 (Actual); Status verified 2023-05

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: Parallel intervention study design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Miffy intervention (Experimental): story of miffy, rewards based on colour they ate
  Interventions: Behavioral: Miffy
- Reward intervetion (Active Comparator): no story, rewards not assigned to colours
  Interventions: Behavioral: Reward
- Control (No Intervention): no story, no rewards

INTERVENTIONS:
Behavioral: Miffy — A method to stimulate children to try different fruits and vegetables using reward and role modelling
  Arms: Miffy intervention
Behavioral: Reward — Reference method to stimulate children to try fruits and vegetables using reward alone
  Arms: Reward intervetion

SUMMARY:
Fruit and vegetable (F&V) intake among children in western countries is below recommended levels. To increase F&V consumption in children (3-6 years), a novel method is proposed based on the concepts of repetitive taste exposure, role models, and non-food rewards guided by the dietary advice: "Eat the rainbow: go for color!" The aim is to determine the effect of this intervention to stimulate the consumption of color on the willingness to try different fruits and vegetables in 210 children aged 3-7 years old

DETAILED DESCRIPTION:
Rationale: A diet rich in fruits and vegetables (F&V) has many health benefits in early childhood. Nevertheless, F&V intake among children in western countries is below recommended levels. To increase F&V consumption in children (3-6 years), a novel method is proposed based on the concepts of repetitive taste exposure, role models, and non-food rewards guided by the dietary advice: "Eat the rainbow: go for color!" Objective: To determine the effect of a modeling- and reward-based intervention to stimulate the consumption of color on the willingness to try different fruits and vegetables in children aged 3-7 years old.

Study design: The study follows a parallel study design. All participants will participate in a baseline session after which they are exposed to a color intervention, a reference intervention, or a control session. Each of the three conditions will be randomly assigned to one of the groups (classrooms) in the participating preschools.

Intervention: The color intervention group listens to a story of Miffy who eats vegetables and fruits in all colors of the rainbow. Afterward, subjects are invited to taste different F&Vs. They are rewarded with a sticker for each color they have eaten. The reference intervention group does not listen to a story and is given a sticker for each type of F&V they have eaten. In the control session, the children are invited to eat F&Vs without any introduction story or reward.

Main study parameters/endpoints: The number of pieces of F&Vs and the number of different types of F&Vs selected, tried, and consumed by the children.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: The study is non-therapeutic to the subjects. No immediate benefits for the subjects are expected from participation in this study, and the risk associated with participation can be considered negligible. In terms of time, the subject's burden is as follows: 30 minutes for the questionnaires prior to the intervention sessions for the caregiver and 15 minutes for the child; 30 minutes for each of the two intervention sessions, however, this coincides with the regular morning break of the children and therefore does not cost extra time, and lastly, 15 minutes for the questionnaire after the intervention sessions for both the child and the caregiver. In total, the time burden amounts to 45 minutes for the participating caregiver and 1 hour and 30 minutes for the participating child.

ELIGIBILITY:
Inclusion Criteria:

* Children in early childhood education and in the first year of primary school within the age range of 3-7.
* Both caregivers as well as the child are willing to comply to the study procedure;

Exclusion Criteria:

* Children who have any allergies or intolerances to the fruits and vegetables used in the study;
* Not willing to eat the test foods because of eating habits or beliefs as indicated by parent or caregiver;

Ages: 3 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 210 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-05-31 (Estimated); Study Completion 2023-05-31 (Estimated)

PRIMARY OUTCOMES:
Change in Willingness to try between | Two sessions (30 minuntes) in two weeks
  Children's' willingness to try pieces of fruit and vegetables is measured in three levels. Children can either eat the study foods or try the study foods:
  A study food is considered as eaten when:
  • The piece of food is completely swallowed by the child;
  A study food is considered as tried when:
  * The piece of food has entered the mouth, but is spit out again;
  * The piece of food is eaten and swallowed, but only partly; The measures are taken by counting the number of pieces of F&V, each of around 30 grams.
  Change in willingness to try is taken between the baseline session (week 1) and the intervention session (week 2)

CONTACTS AND LOCATIONS:
Overall Officials: Guido Camps, Principal Investigator — Wageningen University, Division of Human Nutrition and Health
Locations (1):
- Wageningen University and Research, Wageningen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided